CLINICAL TRIAL: NCT03630263
Title: Impact of Diet in Shaping Gastric Response and RER in Adults From Rural Africa and Urban USA
Brief Title: This Study Assessed the Impact of Diet on Gastric Emptying Time and Metabolic Flexibility
Acronym: IODC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Distinguished Professor of Food Science; Roy L. Whistler Chair, Purdue University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-2019-206
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior
Keywords: Gastric emptying; Postprandial blood glucose
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Repeated measures ANOVA, within factors.
Who Masked: Participant
Masking Description: Participants will be provided with a sample that doesn't contain starch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raw Corn Starch (Experimental): Vehicle (apple sauce) will be spiked with 30 g of slowly digestible carbohydrate (raw corn starch)
  Interventions: Other: Raw Corn Starch
- No Raw Corn Starch (Placebo Comparator): Vehicle (apple sauce) will not be spiked with 30 g of slowly digestible carbohydrate (raw corn starch)
  Interventions: Other: No Raw Corn Starch

INTERVENTIONS:
Other: Raw Corn Starch — Raw corn starch (30 g) will be added to 200 g of applesauce and served to participants, gastric emptying rate, and postprandial glucose will be measured.
  Arms: Raw Corn Starch
Other: No Raw Corn Starch — 200 g of applesauce will be consumed and gastric emptying rate, and postprandial glucose will be measured.
  Arms: No Raw Corn Starch

SUMMARY:
Consumption of slowly digestible carbohydrates can elicit higher satiety feeling compared to rapidly digestible carbohydrates, however not all individuals respond the same. The physiological mechanism that accounts for the satiety effect and the lack of consistency among subjects is not fully understood. The overall aim of this research is to determine if consumption of slow digestible carbohydrates can induce non-responding subjects (i.e., with rapid gastric emptying) to activate the ileal brake and delay rate of gastric emptying.

DETAILED DESCRIPTION:
The purpose of this study is to understand how diet may affect carbohydrate digestion, gastric emptying time and overall health. The investigators will be recruiting 32 volunteers for this study. To be eligible for this study, you need to be between 18 and 50 years old, have a normal Body Mass Index, have a normal fasting blood glucose level, be free of any gastrointestinal diseases, diabetes, cardiovascular diseases, be free of wheat allergens, gluten intolerance or sensitivities, and allergy to millet, and not be pregnant or nursing. If you have any questions about the criteria, please ask the person consenting you.

In this study, participants will consume two test meals at different times to assess gastric emptying times. Test meals will consist of either corn starch (30 g) or pregelatinized (DE-1 Maltodextrin) starch in applesauce (200 g) with xanthan gum (0.2 g) to equalize viscosity. Ingredients will be mixed immediately before consumption. For assessment of gastric emptying time, we will use a non-invasive 13C-labeled octanoic acid breath test. In our proposed procedure, 13C octanoic acid will be added to test meals, and breath samples will be taken before and after ingestion up to 4 hours. Breath samples will be collected every 15 minutes for first 2 hours and every 30 minutes for the next 2 hours. Participants will breathe into 300 mL bags and their content will be evaluated for [13C] using a 13CO2 Urea Breath Analyzer POCone (Otsuka Electronics Co, Ltd, Osaka, Japan) as measures of gastric emptying. We have used the labeled substrate and breath collection methods in our lab under previously approved IRB protocols at Purdue University (IRB Protocols #1102010450, #1104010761, #1209012595, #1405014904, and #1502015807, #1611018484, #1706019377. In addition, before, during, and after each session, subjects will also be asked to fill out a short questionnaire with questions regarding your hunger and fullness at those times. Test meals will be prepared in the university with trained personnel. All the ingredients will be purchased from approved food manufacturers.

During testing days participants will be required to stay in the laboratory. Testing day sessions will last about 4 hours. The day prior testing, participants will be provided a standard meal but are not required to stay.

For assessment of diet composition, three 24-hour dietary recalls will be used. Participants will be called on three different days. During these sessions, participants will be asked to recount quantity and types of foods consumed throughout the day, including two weekdays and one weekend day, to form a comprehensive picture of their dietary habits. Dietary data will be collected and stored using no personally identifiable information.

The purpose of this study is to evaluate the continuous effect of slowly digestible carbohydrates consumption on gastric emptying and its potential health benefits.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25.0 kg/m2
* 18 - 50 years
* Normal fasting blood glucose

Exclusion Criteria:

* History of gastrointestinal disease
* Diabetes
* Pregnant and nursing women
* Wheat and/or gluten allergies or sensitivities
* Allergy to specific sources of slowly digestible carbohydrates

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time | Acute measurement of gastric emptying (4 hours post test meal consumption)
  13C octanoid acid labeled
Metabolic fuel utilization | Acute measures (2 hours post test meal consumption)
  Measured using RER with Lumen

SECONDARY OUTCOMES:
Self reported satiety scores | Acute measurement of satiety or hunger scores (4 hours post test meal consumption)
  Hunger and fullness scores using a 10 cm scale (0=weakest feeling of hunger or fullness; 10=highest or strongest feeling of hunger or fullness)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R Hamaker, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University Lyles Porter Room 1144, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No